CLINICAL TRIAL: NCT01552252
Title: Development and Evaluation of a Low Erosive Apple Juice Drink With Phosphoryl Oligosaccharides of Calcium (POs-Ca)
Brief Title: Evaluation of an Apple Juice Drink With POs-Ca
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hitomi Mita (Other)
Responsible Party: Sponsor-Investigator, Hitomi Mita, Development and Evaluation of a Low Erosive Apple Juice Drink with Phosphoryl Oligosaccharides of Calcium., Tokyo Medical and Dental University
Organization: Tokyo Medical and Dental University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: POs-Ca02
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Food Preferences
Keywords: POs-Ca; calcium additives; drink
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- 0% POs-Ca (Placebo Comparator)
  Interventions: Dietary Supplement: apple juice
- 0.5% POs-Ca (Active Comparator)
  Interventions: Dietary Supplement: apple juice with 0.5% POs-Ca
- 1% POs-Ca (Active Comparator)
  Interventions: Dietary Supplement: apple juice with 1% POs-Ca
- 1.5% POs-Ca (Active Comparator)
  Interventions: Dietary Supplement: apple juice with 1.5% POs-Ca
- 2% POs-Ca (Active Comparator)
  Interventions: Dietary Supplement: apple juice with 2% POs-Ca

INTERVENTIONS:
Dietary Supplement: apple juice — unaltered(0% POs-Ca) commercially available apple juice
  Arms: 0% POs-Ca
Dietary Supplement: apple juice with 0.5% POs-Ca — Phosphoryl Oligosaccharides of Calcium (POs-Ca) in the form of powder was added at concentrations of 0.5% by weight to a commercially available apple juice
  Arms: 0.5% POs-Ca
Dietary Supplement: apple juice with 1% POs-Ca — Phosphoryl Oligosaccharides of Calcium (POs-Ca) in the form of powder was added at concentrations of 1% by weight to a commercially available apple juice
  Arms: 1% POs-Ca
Dietary Supplement: apple juice with 1.5% POs-Ca — Phosphoryl Oligosaccharides of Calcium (POs-Ca) in the form of powder was added at concentrations of 1.5% by weight to a commercially available apple juice
  Arms: 1.5% POs-Ca
Dietary Supplement: apple juice with 2% POs-Ca — Phosphoryl Oligosaccharides of Calcium (POs-Ca) in the form of powder was added at concentrations of 2% by weight to a commercially available apple juice
  Arms: 2% POs-Ca

SUMMARY:
The null hypothesis tested was that there are no differences in the taste palatability of the apple juices before and after adding POs-Ca.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects
* No eating or drinking within 30 minutes before the start time of the trials
* No tooth brushing within 30 minutes before the start time of the trials

Exclusion Criteria:

* apple hypersensibility

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of taste palatability | At time when the subjects have finished drinking, an expected average of 10 minutes
  Tasters were first asked to drink the unaltered (0% POs-Ca) juice, to get familiar with the taste.
  After that they drank each of the 5 juices in a random order, and evaluated the taste by marking an analogue scale ranging from 0 to 100 which was printed horizontally on a sheet of paper.

CONTACTS AND LOCATIONS:
Overall Officials: Hitomi Mita, Principal Investigator — Tokyo Medical and Dental University